CLINICAL TRIAL: NCT07347574
Title: NeuroCare Community Project: A Community Based Prospective Observational Study for Early Alzheimer's Detection in Hong Kong
Brief Title: NeuroCare Community Project: A Community Based Prospective Observational Study for Early Alzheimer's Detection in HK
Status: Not yet recruiting | Type: Observational
Sponsor: Hong Kong University of Science and Technology (Other)
Collaborators: Hong Kong Center for Neurodegenerative Diseases (Other); Tung Wah College (Other)
Responsible Party: Principal Investigator, Hiu Yi Wong, Research Assistant Professor, Hong Kong University of Science and Technology
Other Study IDs: HREP-2025-0390
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: AD - Alzheimer's Disease; Mild Cognitive Impairment; Normal Cognition; Dementia
Keywords: Alzheimer's disease; PET imaging; MR imaging; Biomarker; Amyloid
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitively normal (CN): Participants with normal cognition
  Interventions: Other: Observational
- Mild cognitive impairment (MCI): Participants with MCI
  Interventions: Other: Observational
- Dementia: Participants with dementia
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Clinical profile, blood collection, cognitive assessment, MRI and PET imaging

SUMMARY:
Population aging is reshaping societal dynamics and presents significant global challenges. By 2050, it is projected that 1.6 billion people worldwide will be over the age of 65. Given that aging is the primary risk factor for many common chronic diseases, reducing the burden of age-related illnesses and promoting healthy aging have become critical public health priorities. Notably, Hong Kong has one of the largest proportions of elderly and the highest life expectancy in the world. Dementia, particularly Alzheimer's disease (AD), is a multifaceted condition influenced by both biological and behavioral factors. There is a paucity of robust, community-based prospective data in ethnic Chinese populations that integrate clinical and cognitive measures with objective biomarkers and neuroimaging, especially at earlier stages such as mild cognitive impairment (MCI) and early AD. This community-based project aims to establish a cohort of elderly in Hong Kong, with longitudinal follow-up for 2-3 years. A key strength of this research is the incorporation of a panel of blood biomarkers, which will provide a less invasive and more affordable screening tool to identify Alzheimer's disease at a much earlier stage in the community. Additionally, through benchmark with MRI and PET imaging gold standard, these biomarkers have the potential to predict the conversion risk 1) from clinically normal to mild cognitive impairment and Alzheimer's disease (AD dementia); 2) from clinically MCI to Alzheimer's disease (MCI-AD dementia) or remain static; and differentiate non-AD dementia from Alzheimer's disease (dementia-AD). Collectively, these data will facilitate monitoring of aging processes and cognitive decline, help to identify candidate modifiable factors associated with resilience, and generate a de-identified, Chinese-specific resource to advance healthy aging in Hong Kong.

DETAILED DESCRIPTION:
Introduction Population aging is a major global challenge with estimated 1.6 billion people will be over 65 by 2050. Aging is the main risk factor for many chronic diseases, including Alzheimer's disease (AD). Hong Kong features one of the world's largest proportions of older adults and highest life expectancy and therefore, Hong Kong will face a particular heavy burden on caring of elderly citizens with dementia. Hence, to better planning for caring the aging population within the community, there is a need for robust, community-based data integrating clinical, cognitive, biomarker, and neuroimaging metrics in ethnic Chinese populations. Research Objectives

* Compare validity of clinical assessments, clinical diagnoses, and blood biomarker panels for identifying clinically normal, MCI, and AD using MRI scan and PET imaging as gold standard in a community-based setting.
* Validate blood biomarker panels for predicting conversion from clinically normal to MCI-AD, AD, non-AD MCI/dementia, and MCI to AD/non-AD dementia.
* Explore novel blood and imaging biomarkers for AD diagnosis and progression. Study Design Prospective, community-based cohort study lasting for 5-year duration and expected average 2-3 years longitudinal follow-up for participants.
* Pre-screening of 6,000 community-dwelling elderly at community centers (5-min MoCA, no consent required).
* Enrollment of ~2,500 participants for cross-sectional cohort with informed consent.
* Participants selection and down select as detailed in next section. Participants will undergo clinical, cognitive, and functional assessments; demographic and clinical data collected at local centers.
* Blood sampling by research personnel (HKUST, HKCeND, TWC) with fasting blood processed, analyzed, and stored at HKUST/HKCeND.
* Proteomic results used to stratify participants into low, intermediate, or high risk; imaging follow-up based on stratification. Setting
* Recruitment at district-level community centers for elderly across Hong Kong.
* Centers act as support hubs for healthy aging and provide access to a representative sample.
* Collaboration with Tung Wah College and Tung Wah Group of Hospitals' network. Participant Selection and Down-Selection via Multi-Stage Protocol
* Target: Community-dwelling older adults (Han Chinese, age 60-75) identified through community centers.
* Stage 1 - Brief cognitive screening: 6,000 screened via MoCA-5min; subgroup assignment by percentile (dementia: <2%, mild cognitive impairment (MCI): 2-16%, cognitively normal (CN): >16%).
* Stage 2 - Cross-sectional cohort: 2,500 enrolled, informed consent, clinical and physical assessments, blood tests, clinical diagnosis (DSM-IV). Distribution of subgroups selected: dementia 14%, MCI 43%, and CN 43%.
* Stage 3 - Proteomic sub-cohort: 750 selected for plasma proteomics (21- protein panel + pTau217) and stratified by proteomic score (negative < 21, intermediate 21-52, positive > 52).
* Stage 4 - Imaging sub-cohort: 350 selected for advanced imaging (MRI, amyloid PET) based on clinical diagnosis and proteomic result. All assessments repeated at follow-up for longitudinal monitoring. Variables and Measurement
* Brief Cognitive Function: MoCA-5min: Memory, attention, language, abstraction, orientation.
* Demographics: Age, sex, ethnicity, marital status, family history, education, socio-economic status, occupation.
* Anthropometrics: Height (stadiometer), weight (calibrated scale), BMI calculation.
* Cardiovascular Health: BP, pulse (automated monitor).
* Clinical Assessment Battery: MoCA (full), ADL, iADL, FRAIL, PHQ-9, MBIS.
* Clinical Diagnosis: NIA-AA criteria, applied by registered physicians.
* Blood Tests: 1) Chemistry: Liver, kidney, bone/muscle enzymes, lipids, glucose; 2) Haematology: CBC; 3) Proteomics: Olink, Simoa, Fujirebio, Alamar Biosciences platforms for plasma protein profiling; 4) Genomics (optional): Whole-genome sequencing, methylation arrays, RNA-seq for AD risk loci and gene expression.
* Amyloid/Tau PET and MRI Brain Imaging: PET: Gold standard for amyloid/ tau detection; MRI for structural changes and regional volumetrics.
* Imaging repeated at 2-3 years follow-up for longitudinal assessment.

ELIGIBILITY:
Inclusion Criteria:

* Mentally capable of providing informed consent, with or without an informant present
* Willing and able to undergo blood draw and complete study related assessments; willing to be contacted for follow-up

Exclusion Criteria:

* Lacks capacity to consent even with an informant present
* Refuses or is unable to provide blood samples or complete essential assessments
* Currently enrolled in another clinical trial that could interfere with this study
* Known illness that prevents longitudinal follow up or uncontrolled medical illness such as neurodevelopmental disorder, neurodegenerative disease, epilepsy, central nervous system infection, neuroinflammatory diseases, brain tumor, cerebrovascular diseases, history of major psychiatric illness, history of major head injury with altered consciousness, sexually transmitted disease including HIV and syphilis, visual and auditory disability, history of alcohol dependence, substance use disorder, systemic autoimmune diseases such as systemic lupus erythematosus and rheumatoid arthritis, or malignancy.
* Active delirium or evidence of reversible/secondary causes of cognitive impairment (e.g., vitamin B12 deficiency, hypothyroidism) until treated/ stabilized

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community elderly dwellings
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood biomarker (baseline) | Baseline
  Blood-based biomarkers provide a minimally invasive approach for detecting Alzheimer's disease-related pathology and for monitoring disease progression. Peripheral blood will be analyzed for a core panel that includes p tau217 and a multiplex 21 protein panel, with results generated under predefined quality control specifications.
Follow up blood biomarker | 24 to 36 months after baseline
  Proportion of longitudinally selected participants who complete the repeat fasting blood collection; report completion rate and reasons for non-completion.

SECONDARY OUTCOMES:
Change in MoCA from baseline to follow-up | Baseline to approximately 24-36 months
  Montreal Cognitive Assessment (MoCA), total score 0-30 (higher scores indicate better cognitive function; lower scores indicate worse function); mean change in MoCA total score is calculated based on the difference between MoCA scores at baseline and follow-up visits
Time to cognitive progression | Baseline to approximately 24-36 months
  Time from baseline to clinically adjudicated progression, defined as CN to MCI or dementia, or MCI to dementia, assessed over up to 36 months.
Multimodal imaging data collection | Baseline (PET/MRI within 3-6 months of baseline blood) and repeat at approximately 24-36 months
  Proportion of invited imaging-subset participants who complete planned baseline MRI and amyloid/tau PET according to protocol; repeat completion rate reported at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ip, PhD, Principal Investigator — Hong Kong University of Science and Technology
Locations (1):
- Hong Kong University of Science and Technology, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang Y, Zhou X, Ip FC, Chan P, Chen Y, Lai NCH, Cheung K, Lo RMN, Tong EPS, Wong BWY, Chan ALT, Mok VCT, Kwok TCY, Mok KY, Hardy J, Zetterberg H, Fu AKY, Ip NY. Large-scale plasma proteomic profiling identifies a high-performance biomarker panel for Alzheimer's disease screening and staging. Alzheimers Dement. 2022 Jan;18(1):88-102. doi: 10.1002/alz.12369. Epub 2021 May 25. PMID 34032364
- [Background] Jiang Y, Uhm H, Ip FC, Ouyang L, Lo RMN, Cheng EYL, Cao X, Tan CMC, Law BCH, Ortiz-Romero P, Puig-Pijoan A, Fernandez-Lebrero A, Contador J, Mok KY, Hardy J, Kwok TCY, Mok VCT, Suarez-Calvet M, Zetterberg H, Fu AKY, Ip NY. A blood-based multi-pathway biomarker assay for early detection and staging of Alzheimer's disease across ethnic groups. Alzheimers Dement. 2024 Mar;20(3):2000-2015. doi: 10.1002/alz.13676. Epub 2024 Jan 6. PMID 38183344